CLINICAL TRIAL: NCT02014168
Title: A Phase I Study to Determine the Safety and Immunogenicity of Co-administration of the Candidate Influenza Vaccine MVA-NP+M1 and the Viroflu® Seasonal Influenza Vaccine
Brief Title: Safety and Immunogenicity of Co-administration of Candidate Influenza Vaccine MVA-NP+M1 and Viroflu® Seasonal Influenza Vaccine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Futility
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLU006; 2013-003569-32 (EudraCT Number)
Record Dates: First submitted 2013-11-08; First posted 2013-12-18 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viroflu® and MVA-NP+M1 (Experimental): 1 dose (0.5ml) of Viroflu® and 1 dose of 1.5 x10^8 pfu MVA-NP+M1 intramuscularly into the vastus lateralis muscle on day 0. The vaccines will be given side by side, with MVA NP+M1 being given immediately after the seasonal influenza vaccine.
  Interventions: Biological: Viroflu® and MVA-NP+M1
- Viroflu® and saline placebo (Placebo Comparator): 1 dose (0.5ml) of Viroflu® and 1 dose of a 0.9% saline placebo injected intramuscularly into the vastus lateralis muscle on day 0. The placebo will be administered immediately after the seasonal influenza vaccine.
  Interventions: Biological: Viroflu® and saline placebo

INTERVENTIONS:
Biological: Viroflu® and MVA-NP+M1 — 2013-2014 season Viroflu, manufactured by Crucell. Contains 15 microgrammes of haemagglutinin (HA) from an H1N1 subtype influenza A virus, an H3N2 subtype influenza A virus and an influenza B virus per 0.5 ml dose.
  MVA-NP+M1 manufactured by by IDT Biologika GmbH, Germany. Each vial of MVA-NP+M1 contains 700 microlitres volume at a concentration of 1.3 x108 pfu/ml in 10mM Tris buffer. The dose of MVA-NP+M1 to be used in this study will be 1.5 x108 pfu.
  Other Names: Viroflu®; Viroflu; MVA-NP+M1
  Arms: Viroflu® and MVA-NP+M1
Biological: Viroflu® and saline placebo — 2013-2014 season Viroflu, manufactured by Crucell. Contains 15 microgrammes of haemagglutinin (HA) from an H1N1 subtype influenza A virus, an H3N2 subtype influenza A virus and an influenza B virus per 0.5 ml dose.
  0.9% saline placebo.
  Other Names: Viroflu®; Viroflu
  Arms: Viroflu® and saline placebo

SUMMARY:
This is a single blinded placebo controlled phase I study, to assess the safety and immunogenicity of co-administration of the candidate influenza vaccine MVA-NP+M1 with the Viroflu® seasonal influenza vaccine. All volunteers recruited will be healthy adults aged 18 and over.

DETAILED DESCRIPTION:
This study is designed to test the safety and effectiveness of a combination of two vaccines for influenza. One of these vaccines will be the seasonal influenza vaccine 'Viroflu' ('Inflexal V'). The second will be an investigational viral vectored vaccine called MVA NP+M1. The rationale for combining these two vaccines is that they work differently and that by combining the two vaccines, stronger and broader immune responses may be produced.

The MVA NP+M1 vaccine has been evaluated in five previous clinical trials. In total, over 80 volunteers have received this vaccine. There have been no vaccine related serious adverse events. Higher doses of MVA NP+M1 are more reactogenic, however at the dose to be used in this study the majority of adverse events are mild.

20 volunteers will be recruited in this study. They will all be adults over the age of 18. Volunteers will be assigned to one of two groups. Volunteers in group 1 will receive Viroflu, followed by a dose of MVA NP+M1. Volunteers in group 2 will receive Viroflu followed by a placebo injection (saline). Volunteers will be blinded so that they do not know which group they have been allocated to and will be asked to complete diary cards listing any adverse events after vaccination.

Vaccinations will be administered into the thigh as the deltoid muscle is not normally large enough to accept two intramuscular injections.

Volunteers will followed up for 6 months in total. Two days after vaccination they will receive a telephone call from one of the clinical team. They will then attend three follow up visits (at weeks 1, 3 and 26). At each visit, volunteers will have blood tests taken and will be questioned about any adverse events they may have experienced.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 years and over
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For heterosexual, pre-menopausal females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day of vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational influenza vaccine, or any other investigational vaccine likely to impact on interpretation of the trial data.
* Receipt of the 2013/14 seasonal influenza vaccine prior to entering the study.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled/topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Any history of anaphylaxis in reaction to vaccination
* Recent treatment for cancer (except basal cell carcinoma and cervical carcinoma in situ)
* History of a serious psychiatric condition
* Suspected or known current injecting drug or alcohol abuse (as defined by an alcohol intake of greater than 42 units every week)
* Seropositive for hepatitis B surface (HBsAg) or hepatitis C virus (antibodies to HCV) For pre-menopausal females, pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other significant disease, disorder or finding (including blood test results), which, in the opinion of the Investigators, would either put the volunteer at risk because of participation in the study, or may influence the result of the study.
* No response / confirmation from GP regarding previous medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cellular immune response generated by co-administration of MVA-NP+M1 and the Viroflu® seasonal influenza vaccine | 26 weeks
  Interferon-gamma ELISpot will be used as a marker of cell-mediated immunity.
Humoral immune response generated by co-administration of MVA-NP+M1 and the Viroflu® seasonal influenza vaccine | 26 weeks
  Humoral response will be measured by HI titre, ELISA, or neutralising antibody assay.

SECONDARY OUTCOMES:
Safety of co-administration of MVA-NP+M1 and the Viroflu® seasonal influenza vaccine | Participants will be followed for the duration of the study, an expected average of 6 months
  Data pertaining to adverse events will be actively and passively collected; the data will be presented according to frequency, severity and duration of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V S Hill, DPhil FRCP, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, Oxfordshire, United Kingdom